CLINICAL TRIAL: NCT00978744
Title: Evaluation of a Regional Electronic Health Information Exchange's Clinical Health Record
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Shared Health, Chattanooga, TN (Unknown)
Responsible Party: Principal Investigator, Jeffrey Rothschild, MD, Hospitalist, Brigham and Women's Hospital
Other Study IDs: 2007-P-002256/1; BWH
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Impact of Health Information Exchange on Patient Care; (Focus on Diabetes, Asthma, Hypertension, CHF, COPD, CAD,; Gastroenteritis, Seizures, and Bacterial Pneumonia)
Keywords: Clinical Health Record; Computerized Decision Support; Patient Safety; Resource Utilization
MeSH Terms: conditions — Diabetes Mellitus; Asthma; Hypertension; Heart Failure; Pulmonary Disease, Chronic Obstructive; Gastroenteritis; Seizures; Pneumonia, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The Shared Health CHR™ (Clinical Health Record) offers point-of-care clinical reporting and decision support based primarily on patient claims data aggregated across various health care settings, and is one example of the types of health information data exchange efforts being implemented across the country. This study will evaluate how the CHR is used and its clinical and financial impact to better understand the CHR's value, and to identify opportunities to enhance the system to support patient care and practice efficiency. In addition, the results from this study will help to inform the national debate about the effectiveness of these types of tools to maximize patient quality of care, patient safety, and practice efficiency.

DETAILED DESCRIPTION:
Missing information at the point of care is frustrating for both physicians and patients and can lead to unnecessary tests or suboptimal or even inappropriate and potentially harmful treatment. In addition to the risks of poorer quality of care, this fragmentation of incomplete or unavailable clinical data may result in increased costs to the healthcare system. Patient health records, when electronically shared across a spectrum of patient care settings, offer the possibility of improving healthcare outcomes, including patient safety and quality of care, and increasing efficiency, as well as cost-effectiveness.

This overall study will consist of two analyses. First, we will conduct a before-and-after, or pre-post study. The clinical practices consenting to participate will serve as their own controls during the baseline period. During the baseline period for which data will be retrospectively captured, physicians will have been conducting "business as usual" without the use of the CHR. The intervention will consist of participants accessing CHR to assist with medical decisions and patient care. Secondly, we will conduct a concurrent matched cohort comparison of patients within practices. We will compare outcomes and gaps in care for patients whose care is associated with very frequent CHR use and less frequent CHR use to matched control patients whose care is not associated with CHR use.

Safety, quality, and cost outcomes will be compared using the two described approaches. First, we will compare outcomes and gaps in care for the intervention patients whose care involved active CHR use in the intervention period to the care these same patients received during the baseline periods (pre/post analyses). Secondly, we will compare outcomes and gaps in care of the intervention active patients, both super-active and less active, to the matched control patients whose care during the study did not involve any CHR use during the intervention period (matched cohort analysis).

In order to study the relationship of CHR use to clinical, financial, and office efficiency outcomes within the study's timeline, we will limit our study to pre-existing patients and new patients who have had at least one encounter during the study period. Hospital admission data will also be analyzed as part of the cost and outcomes analysis.

We plan to study the effects of CHR on several conditions among the AHRQ's Ambulatory Care Sensitive (ACS) Conditions. We will study conditions that are common, high-risk, and resource dependent where clinical management may be improved with access to a CHR including chronic obstructive pulmonary disease/asthma, congestive heart failure, angina/coronary artery disease, and diabetes mellitus. In addition, other conditions determined to be of value in evaluating the impact of the CHR may be added, or may replace some of the existing conditions. These conditions will be chosen based on our early work in the study once we learn more about the number of eligible patients and the numbers of clinical interactions. The new conditions, yet to be determined, may also include non-chronic, or acute, diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be primary care clinicians (nurse practitioner, physician assistant, or physician) who have registered to use the CHR at a practice that is enrolled in the study.

Exclusion Criteria:

* Specialty clinicians are excluded.
* Primary care clinicians who have not registered to use the CHR at an enrolled practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are not being enrolled as subjects; their deidentified data will be reviewed only if their associated physicians and practices are participating as subjects in the study. Physicians, staff, and patients within the study population are representative of the practices we are going to study. Patients' data will be included in the intervention study to the extent that they are part of Shared Health's CHR system, are receiving care at one of the selected practices, and meet eligibility requirements.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2008-12; Primary Completion 2012-01 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Gaps in care; compliance with quality measures | 2008 baseline, 2009-2010 intervention
  Data are collected from Shared Health about the outcome measures for baseline period (calendar year 2008) and for the intervention period which is 2009-2010 phased across the participating practices depending on when they implemented the clinical health record.

SECONDARY OUTCOMES:
Costs of care | 2008 baseline, 2009-2010 intervention
  Costs of care are being evaluated for the baseline period of 2008 and for the intervention period of 2009-2010 which is phased across participating practices depending on when they implemented the clinical health record.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rothschild, MD, Principal Investigator — Brigham and Women's Hospital